CLINICAL TRIAL: NCT03304184
Title: The Role of Biodentine in Class V Dental Lesions on Oral Health Related Quality of Life
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elizabeth Van Tubergen, Clinical Assistant professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00111890
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Quality of Life; Cervical Abrasion

STUDY DESIGN:
Intervention Model Description: One group will be treated with a tooth colored filling that will be placed near the gum line. The second group will be treated with a white colored filling that will be placed near the gum line.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Photac-fil (Placebo Comparator): Participants will have a restoration placed with photac-fil in the lesion near the gum line.
  Interventions: Device: Photac-fil
- Biodentine (Experimental): Participants will have a restoration placed with Biodentine in the lesion near the gum line.
  Interventions: Device: Biodentine

INTERVENTIONS:
Device: Photac-fil — Application of a tooth colored filling in a non-cavitated dental lesion.
  Other Names: Resin modified glass ionomer
  Arms: Photac-fil
Device: Biodentine — Application of a white colored filling in a non-cavitated dental lesion.
  Arms: Biodentine

SUMMARY:
The study will compare two different dental materials on dental lesions near the gum line that cause chronic pain on oral health related quality of life.

DETAILED DESCRIPTION:
The study will compare two different dental materials on dental lesions near the gum line. One of the materials is tooth colored and the other material is white but both materials use different mechanisms to attach to the teeth and may have different outcomes. The study will determine if one material is more effective in relieving chronic pain. In addition, we will evaluate changes in oral health related quality of life after the placement of the two different dental materials.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18-64
* Chief complaint associated with pain from cold or hot
* Chronic sensitivity associated with supragingival lesions
* Pain not associated with decay
* Fluent in English and able to read English at a 6th grade level
* Pulpal response <40 via pulp tester
* Active salivary flow from palpation of parotid and submandibular glands
* Patients self reporting pain over 6/10 in the past week and/or the past 2 months

Exclusion Criteria:

* Pregnant women
* Patients taking benzodiazepines, narcotics and multiple antidepressants for pain management not associated with the oral cavity
* Unexplained dry mouth
* Patients taking two or more medications associated with dry mouth
* Pulpal response >40 via pulp tester
* Patients requiring treatment for more than 5 decayed sites, periodontal disease and root canal therapy
* Complicated medical history (>4 concurrent treatment for systemic diseases)
* Lesion >1mm below the gum line

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dental School, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Photac-fil | Biodentine
Started | 15 | 9
Completed (Participants that completed all of the survey questions over a 3 month period.) | 14 | 7
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photac-fil | Biodentine | Total
Number analyzed (Participants) | 15 | 9 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 9 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 8 | 21
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 7 | 7 | 14
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Global Base Changes of Pain
Description: A one survey description detailing the changes in pain over time based on the following scale:
  1. -No change (or condition has gotten worse)
  2. -Almost the same, hardly any change at all
  3. -A little better, but no noticeable change
  4. -Somewhat better, but the change has not made any real difference
  5. -Moderately better, and a slight but noticeable change
  6. -Better and a definite improvement that has made a real and worthwhile difference
  7. -A great deal better and a considerable improvement that has made all the difference
Time Frame: baseline, week1, week 2, 3 month follow up
Population: Global Base Changes of pain measured over 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Photac-fil | Biodentine
Number analyzed (Participants) | 15 | 9
units on a scale
  Global base changes-baseline | 3.2 (2.4) | 2.3 (2.1)
  Global base changes-week 1 | 5.9 (1.6) | 4.6 (2.3)
  Global base changes-week 2 | 6.3 (.6) | 4.5 (2.2)
  Global base changes-3 month follow up | 6.4 (.6) | 4.6 (2.4)
Statistical Analysis 1: Comparison: Photac-fil vs Biodentine; Power was limited sample size between the groups a superiority analysis was not able to be completed, so an equivalence test was used; Test type: Equivalence — In this analysis, the null hypothesis was that there was no significant difference in global base changes scores between the two treatment groups (Photac and Biodentine); p = .0001, ANOVA; Mean Difference (Final Values) = 3 — The estimation values were from an average of all values in each arm
Statistical Analysis 2: Comparison: Photac-fil vs Biodentine; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — In this analysis, the null hypothesis was that there was no significant difference in global base changes scores between the two treatment groups (Photac and Biodentine) over timepoints; p = .0005, ANOVA; Mean Difference (Final Values) = 3 — The estimation values were from an average of all values in each arm

2. Primary Outcome: Oral Health Related Quality of Life Using a Survey With 49 Questions
Description: A survey of 49 questions to assess oral health related quality of life. The scale measured 49 questions with a yes (1) or no (0) answers with a possible range of 0-49. The more answers of yes will indicate a higher score on the survey, which describes poorer oral health related quality of life. A lower number reflects better oral health related quality of life. A maximum score of 49 is the worst outcome.
Time Frame: Baseline, week1, week 2, 3 month follow up
Population: OHIP-49 score for Photac group measured over 3 months
Measure: Mean (Standard Deviation); unit: total score
Groups:
- Photac: Participants will have a restoration placed with photac-fil in the lesion near the gum line.
  Photac-fil: Application of a tooth colored filling in a non-cavitated dental lesion.
Arm/Group | Photac | Biodentine
Number analyzed (Participants) | 15 | 9
total score
  Baseline measurement | 11.5 (11.2) | 14.4 (14.6)
  Week 1 measurement | 5.5 (8.1) | 12.7 (18.9)
  Week 2 measurement | 4.5 (6.9) | 7.4 (11.5)
  3 month follow up | 2.6 (5.1) | 4.9 (7.0)
Statistical Analysis 1: Comparison: Photac vs Biodentine; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — In this analysis, the null hypothesis was that there was no significant difference in 49 questions on oral health related quality of life scores between the two treatment groups (Photac and Biodentine); p = .0910, ANOVA — Comparison between two groups for treatment; Mean Difference (Final Values) = 3 — The estimation values were from an average of all values in each arm
Statistical Analysis 2: Comparison: Photac vs Biodentine; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — In this analysis, the null hypothesis was that there was no significant difference in 49 questions on oral health related quality of life scores between the two treatment groups (Photac and Biodentine) over time points; p = .0262, ANOVA — Comparison between the two arms for treatment time points with analysis; Mean Difference (Final Values) = 3 — The estimation values were from an average of all values in each arm

3. Primary Outcome: Brief Pain Inventory
Description: 6 questions were used to measure pain on a sliding scale from 1-100 at each time point. The scale ranged from 1 being no pain and 100 being extreme pain. The higher the number reflects worse the pain compared to a lower number. The maximum range from the participants was 600 (maximum) and the lowest range of 0 for all questions. The data reflects the averaged sum for each time point for all patients in each arm.
Time Frame: Baseline, week1, week 2, 3 month follow up
Population: Brief pain inventory measured over time
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Photac-fil | Biodentine
Number analyzed (Participants) | 15 | 9
score on a scale
  Brief pain inventory score- baseline | 152.4 (106.3) | 192.6 (169.5)
  Brief pain inventory score- week 1 | 103.1 (122.8) | 141.1 (179.1)
  Brief pain inventory score- week 2 | 91 (134.8) | 66.8 (71.7)
  Brief pain inventory score- 3 month recall | 55 (96.4) | 76.8 (122.3)
Statistical Analysis 1: Comparison: Photac-fil vs Biodentine; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — In this analysis, the null hypothesis was that there was no significant difference in brief pain inventory scores between the two treatment groups (Photac and Biodentine) over different time points; p = .0289, ANOVA; Mean Difference (Final Values) = 3 — The estimation values were from an average of all values in each arm

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the first two weeks of the placement of Biodentine as the material debonded from the tooth.
Description: If any of the treatment arms have a deviation as a result of the restoration falling out or debonding, it is not a serious adverse event because the tooth was not prepped prior to the placement of the restoration. This would result in the area of the tooth that lost the restoration going back to the pre-treatment form. This would also not result in any risk of mortality.
Arm/Group | Photac-fil | Biodentine
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/9
Other Adverse Events (participants affected / at risk) | 0/15 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photac-fil (N=15) | Biodentine (N=9)
Debonding of Biodentine from area added (Product Issues) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT03304184/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03304184/ICF_003.pdf